CLINICAL TRIAL: NCT00629694
Title: Adenoidectomy, Myringotomy and Tubes' Insertion vs Adenoidectomy and Myringotomy Alone in Children With Otitis Media With Effusion and Adenoid Hypertrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aghia Sophia Children's Hospital of Athens (Other)
Responsible Party: Principal Investigator, Ioannis Vlastos, MD, Aghia Sophia Children's Hospital of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-01-07
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Otitis Media With Effusion
Keywords: adenoidectomy, myringotomy, tubes insertion, otitis media, adenoid hyperthophy
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media | interventions — Adenoidectomy; Middle Ear Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- A-T (Active Comparator)
  Interventions: Procedure: adenoidectomy, myringotomy, tubes insertion
- A-M (Experimental)
  Interventions: Procedure: A-M

INTERVENTIONS:
Procedure: adenoidectomy, myringotomy, tubes insertion — adenoidectomy, myringotomy and tubes insertion (A-T)against adenoidectomy and myringotomy alone (A-M)
  Arms: A-T
Procedure: A-M — adenoidectomy and myringotomy alone
  Arms: A-M

SUMMARY:
It is not unusual for several children operated for severe adenoid hyperthrophy causing breathing problems to have otitis media with effusion simultaneously. It is unknown whether adenoidectomy, myringotomy and tubes insertion is superior to adenoidectomy and myringotomy alone in terms of otitis media related quality of life and recurrence of otitis media several months after the operation. For this purpose a randomized trial is conducted including children operated for adenoid hyperthrophy and whose otitis media with effusion had caused minimal or no symptoms so far

ELIGIBILITY:
Inclusion Criteria:

* children operated for their adenoid hyperthrophy with an adenoid size of 3 (measured in a scale of 1-3 intraoperatively or from lateral neck x-ray) and otitis media with effusion causing an average air-bone gap of greater than 20db. Children should be otherwise healthy with an ASA score of I and between 3-12 years old of age

Exclusion Criteria:

* other health problems especially related with the condition eg cleft palate

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
OM-6 | one year post operative

SECONDARY OUTCOMES:
tympanogram type B | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis M Vlastos, MD, Principal Investigator — Aghia Sophia Children's Hospital of Athens
Locations (1):
- Department of Otolaryngology-Head and Neck Surgery, Aghia Sophia Children's Hospital of Athens, Athens, Greece